CLINICAL TRIAL: NCT01460667
Title: A Randomized, Double-Blind, Placebo-Controlled, Single Center Study of IV Acetaminophen for the Treatment of Post-Operative Pain After Laparoscopic Roux-en-Y Gastric Bypass Surgery (LRYGBP)
Brief Title: Efficacy of IV Acetaminophen in Acute Post-Operative Pain Control in Laparoscopic Roux-en-Y Gastric Bypass Surgery (LRYGBP) Patients
Acronym: IV APAP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: McLaren Regional Medical Center (Other)
Collaborators: Cadence Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Christina Lee, Study Coordinator, McLaren Regional Medical Center, McLaren Regional Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IV APAP LRYGBP Study
Record Dates: First submitted 2011-10-19; First posted 2011-10-27 (Estimated); Last update posted 2011-10-27 (Estimated); Status verified 2011-10

CONDITIONS: Morbid Obesity
Keywords: Laparoscopic Roux-en-Y Gastric Bypass; Post-Operative Pain; IV Acetaminophen; Post-Operative Nausea and Vomiting
MeSH Terms: conditions — Obesity, Morbid; Pain, Postoperative; Vomiting | interventions — Acetaminophen; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IV acetaminophen (Active Comparator)
  Interventions: Drug: IV acetaminophen
- IV 0.9% normal saline (Placebo Comparator)
  Interventions: Drug: IV normal saline

INTERVENTIONS:
Drug: IV acetaminophen — IV acetaminophen 1000 mg (100 mL) every 6 hours over 30 hours
  Arms: IV acetaminophen
Drug: IV normal saline — 0.9% normal saline IV, every 6 hours over 30 hours.
  Arms: IV 0.9% normal saline

SUMMARY:
Laparoscopic Roux-en-Y gastric bypass (LRYGBP) is a common type of surgery in which length of stay and morbidity is intimately associated with post-operative nausea and vomiting (PONV) and recovery of bowel function. Medications most commonly used to control for post-operative pain are opioid medications, whose well known adverse effects include PONV. Currently, no studied adequate alternative to opiates exists for mild-moderate pain relief without the aforementioned risks.

The primary goal for this study is to evaluate the the administration of pre- and post-operative IV acetaminophen to determine if there is in an overall decrease in the use of opioid analgesics by patient controlled analgesia (PCA) and subsequent decrease in subjective PONV leading to sooner return of bowel function, enabling progression to oral intake and decrease in post-operative length of stay.

DETAILED DESCRIPTION:
Opioid use during the post-operative period is a highly effective means of treatment for acute pain, however not without its adverse effects including post-operative nausea, vomiting (PONV), constipation, urinary retention, sedation and respiratory depression. Such factors have been implied in the literature to contribute to prolonged post-operative length of stay, delayed return to diet, return of bowel function and increased incidence of ileus. Alternatively, non-opioids, such as acetaminophen, aspirin, NSAIDs, and selective cyclo-oxygenase-2 inhibitors, can be utilized for acute pain, either alone or in combination with opioids. In the bariatric post-surgical population, NSAIDS both oral and IV (Toradol, Ibuprofen) are not recommended due to their potential bleeding tendency, anti-inflammatory effect, and ulcerogenic effect.

The LRYGBP may be classified as a surgery type associated with mild to moderate post-operative pain. Therefore, the mode of pain relief could directly affect the length of stay. The advent of IV acetaminophen serves as a opportunity to investigate in detail the efficacy of this non-opioid medication in the management of acute pain in the immediate post-operative period without the aforementioned adverse effects as expected from traditional opiate medications. A comprehensive approach to this study includes a prospective, double-blinded, randomized controlled trial of subjects who will undergo LRYGBP and randomized to the study agent (IV acetaminophen) or placebo.

ELIGIBILITY:
Inclusion Criteria:

* patients who are scheduled to undergo laparoscopic Roux-en-Y gastric bypass surgery (LRYGBP) under general anesthesia.
* age 18 to 65 years
* BMI >35
* ASA scores 1,2, or 3
* a negative pregnancy test for female subjects of childbearing age
* ability to read, understand and provide informed consent to the study procedures
* ability to read and understand the use of pain and nausea scales (VAS)

Exclusion Criteria:

* known hypersensitivity to acetaminophen or opioids
* use of opioid or schedule II medications prior to commencement of the study >7 days
* those with chronic pain conditions or significant medical disease requiring pain control
* abnormal liver function (aspartate aminotransferase/alanine aminotransferase/bilirubin > 3X upper limit of normal range, active hepatic disease, clinically significant liver disease, cirrhosis or hepatitis)
* known or suspected alcohol, drug or opiate abuse or dependence; or participation in other clinical study within 30 days of surgery.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Estimated)
Dates: Start 2011-10; Primary Completion 2012-10 (Estimated)

PRIMARY OUTCOMES:
difference in post-operative opiate consumption (PCA) | hourly, 30 hours from first dose of study agent

SECONDARY OUTCOMES:
post-operative subjective pain intensity | every 2 hours, 30 hours from first dose of study agent
post-operative nausea and vomiting (PONV) | every 2 hours, 30 hours from first dose of study agent
time to first post-operative drug administration | up to 30 hours from first dose of study agent
time to return to flatus | up to 30 hours from first dose of study agent
acceptance of rescue medication | up to 30 hours from first dose of study agent
time to first request for rescue medication | up to 30 hours from first dose of study agent
readiness for discharge | up to 72 hours from the first dose of study agent

CONTACTS AND LOCATIONS:
Overall Officials: Christina Lee, B.Sc., Study Director — McLaren Regional Medical Center
Locations (1):
- McLaren Regional Medical Center, Flint, Michigan, United States

REFERENCES:
- [Background] Nguyen NT, Ho HS, Palmer LS, Wolfe BM. A comparison study of laparoscopic versus open gastric bypass for morbid obesity. J Am Coll Surg. 2000 Aug;191(2):149-55; discussion 155-7. doi: 10.1016/s1072-7515(00)00276-3. PMID 10945358
- [Result] Walder B, Schafer M, Henzi I, Tramer MR. Efficacy and safety of patient-controlled opioid analgesia for acute postoperative pain. A quantitative systematic review. Acta Anaesthesiol Scand. 2001 Aug;45(7):795-804. doi: 10.1034/j.1399-6576.2001.045007795.x. PMID 11472277
- [Result] Macario A, Royal MA. A literature review of randomized clinical trials of intravenous acetaminophen (paracetamol) for acute postoperative pain. Pain Pract. 2011 May-Jun;11(3):290-6. doi: 10.1111/j.1533-2500.2010.00426.x. Epub 2010 Nov 28. PMID 21114616
- [Result] Wininger SJ, Miller H, Minkowitz HS, Royal MA, Ang RY, Breitmeyer JB, Singla NK. A randomized, double-blind, placebo-controlled, multicenter, repeat-dose study of two intravenous acetaminophen dosing regimens for the treatment of pain after abdominal laparoscopic surgery. Clin Ther. 2010 Dec;32(14):2348-69. doi: 10.1016/j.clinthera.2010.12.011. PMID 21353105
- [Result] Madan AK, Ternovits CA, Speck KE, Tichansky DS. Inpatient pain medication requirements after laparoscopic gastric bypass. Obes Surg. 2005 Jun-Jul;15(6):778-81. doi: 10.1381/0960892054222812. PMID 15978146